CLINICAL TRIAL: NCT03781843
Title: Effects of Genicular Nerve Block for Patients With Knee Osteoarthritis Who Have Neuropathic or Nociceptive Pain: A Double-Blind, Randomized Controlled Trial
Brief Title: Effects of Genicular Nerve Block in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berrak Tas, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018/42
Record Dates: First submitted 2018-11-27; First posted 2018-12-20 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-12

CONDITIONS: Knee Osteoarthritis
Keywords: Neuropathic Pain; Nerve block; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Neuralgia | interventions — Lidocaine; Sodium Chloride; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Genicular nerve block with lidocaine (Active Comparator): The ultrasound-guided genicular nerve block was performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. Color Doppler was used to identify the arterial structures which serve as landmarks for the corresponding nerves.10 cm 21 G insulated block needle was inserted and aligned with the ultrasound scanning plane. Once satisfactory position of the needle is confirmed, 6 mL of a solution containing 6 mL of 2% lidocaine or 6 mL dextrose or 6 mL saline was slowly injected. Spread of local anesthetic was documented adjacent to the target nerve. This procedure was performed at the site of the three genicular nerves Interventions: Drug: 6 mL 2% lidocaine Procedure: Genicular nerve block
  Interventions: Drug: Genicular nerve block with lidocaine
- Genicular nerve block with saline (Placebo Comparator): The ultrasound-guided genicular nerve block was performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. Color Doppler was used to identify the arterial structures which serve as landmarks for the corresponding nerves.
  10 cm 21 G insulated block needle was inserted and aligned with the ultrasound scanning plane. Once satisfactory position of the needle time is confirmed, 5 mL of a saline was slowly injected. Spread of local anesthetic was documented adjacent to the target nerve. This procedure was performed at the site of the three genicular nerves.
  Interventions:Drug: Saline Procedure: Genicular nerve block
  Interventions: Drug: Genicular nerve block with saline
- Genicular nerve block with dextrose (Placebo Comparator): The ultrasound-guided genicular nerve block was performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. Color Doppler was used to identify the arterial structures which serve as landmarks for the corresponding nerves.
  10 cm 21 G insulated block needle was inserted and aligned with the ultrasound scanning plane. Once satisfactory position of the needle time is confirmed, 5 mL of a dextrose was slowly injected. Spread of local anesthetic was documented adjacent to the target nerve. This procedure was performed at the site of the three genicular nerves.
  Interventions:Drug: Dextrose Procedure: Genicular nerve block
  Interventions: Drug: Genicular nerve block with dextrose

INTERVENTIONS:
Drug: Genicular nerve block with lidocaine — The color doppler ultrasound-guided genicular nerve block at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves.
  Arms: Genicular nerve block with lidocaine
Drug: Genicular nerve block with saline — The color doppler ultrasound-guided genicular nerve block at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves.
  Arms: Genicular nerve block with saline
Drug: Genicular nerve block with dextrose — The color doppler ultrasound-guided genicular nerve block at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves.
  Arms: Genicular nerve block with dextrose

SUMMARY:
Genicular nerve block is a safe and effective therapeutic procedure for intractable pain associated with chronic knee osteoarthritis (OA). There is increasing support for the neuropathic component to the knee OA pain. Investigators proposed that targeting treatment to the underlying pain mechanism can improve pain management in knee OA. There is a debate on injectable solutions used in nerve blocks. Investigators aimed to investigate the efficacy of genicular nerve block and to determine which solution should be appropriate for patients with knee osteoarthritis who have neuropathic or nociceptive pain.

DETAILED DESCRIPTION:
The patients who participated in this study were selected from outpatients who attended our hospital for knee pain. These 90 patients were who matched the following criteria. All patients had knee pain for more than 3 months.

The ultrasound-guided genicular nerve block was performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. Color Doppler was used to identify the arterial structures which serve as landmarks for the corresponding nerves. This method was used to inject a total of 6 mL of lidocaine or 6 mL dextrose or 6 mL saline at 3 separate target sites: the superior lateral, superior medial, and inferior medial genicular nerves.

Pain was evaluated with Analog Analogue Scale (VAS), daily living activities with Western Ontario and McMaster Universities Arthritis Index (WOMAC), maximum distance walked with Lequesne Score, and neuropathic pain was evaluated with painDETECT inquiry form. Outcome measures were assessed at baseline and at 1st, 4th weeks, and 3rd months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* knee pain for more than 3 month.
* radiological tibiofemoral OA (Kellgren-Lawrence grade 2-4 )

Exclusion Criteria:

* acute knee pain, prior knee surgery, other connective tissue diseases that affected the knee, serious neurological or psychiatric disorders, steroid or hyaluronic acid injection therapy during the previous 3 months, sciatic pain, patients with polyneuropathy, anticoagulant medication use, pacemaker use, prior electroacupuncture treatment and physical treatment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-29 (Estimated)

PRIMARY OUTCOMES:
Efficacy of genicular nerve block on neuropathic pain reduction in knee osteoarthritis | 3 months
  Neuropathic pain reduction is measured by painDETECT questionnaire (PD-Q) which consists of 9 items that evaluate pain quality, pattern and radiation. Possible scores range from -1 to 38, with higher scores indicating more neuropathic-like symptoms. Clinical assessments:score ≤12: unlikely neuropathic pain; score 13-18: possibly neuropathic pain, and score ≥19:likely neuropathic pain.
Efficacy of genicular nerve block on nociceptive pain reduction in knee osteoarthritis. | 3 months
  Nociceptive pain reduction is measured by Visual analogue scales (VAS). The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).

SECONDARY OUTCOMES:
Efficacy of genicular nerve block on physical function in knee osteoarthritis. | 6 months
  Physical functional disability is measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC index is a self-administered health questionnaire specifically designed for patients with osteoarthritis of the hip or knee. It consists of 24 multiple-choice items grouped into 3 categories: WOMAC pain, WOMAC stiffness, and WOMAC physical function. The questions are ranked on a 5-point Likert scale (1 point, best result; 5 points, worst result), and the scores are added up for each category. The WOMAC scores from 1 (best) to 5 (worst) points to a system of 0 (worst) to 100 (best) points.
Efficacy of genicular nerve block on walking distance in knee osteoarthritis. | 6 months
  Walking distance with or without walking aids is measured by Lequesne algofunctional index.The Lequesne OA index is a 11-question interview format questionnaire with three sections about pain or discomfort, maximum distance walked and possible necessity of crutches and activities of daily living . The Lequesne OA index is scored as the sum of all questions ranging from 0 to 24. Lower score indicates less dysfunction where 0 = no handicap, 1-4 = mild handicap, 5-7 = moderate handicap, 8-10 = severe handicap, 11-13 = very severe handicap, and ≥14 = extremely severe handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Akpınar, MD, Study Director — FATİH SULTAN MEHMET EDUCATION AND RESEARCH HOSPITAL
Locations (1):
- Fatih Sultan Mehmet Education and Research Hospital, Istanbul, Turkey (Türkiye)